CLINICAL TRIAL: NCT01423760
Title: An Open-label Trial to Collect Long-term Data on Subjects Following Participation in Previous EMD 531444 (L-BLP25 or BLP25 Liposome Vaccine) Clinical Trials
Brief Title: Common Safety Follow-up Trial of Tecemotide (L-BLP25)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is terminated prematurely as the sponsor decided to discontinue program with Tecemotide in NSCLC.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 63325-011
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small Cell Lung Cancer; Multiple Myeloma
Keywords: Vaccine; Stimuvax; Tecemotide; L-BLP25; Non-Small Cell Lung Carcinoma; Multiple Myeloma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Multiple Myeloma | interventions — L-BLP25

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tecemotide (L-BLP25) (Experimental)
  Interventions: Biological: Tecemotide
- Observational (Other)
  Interventions: Other: No intervention

INTERVENTIONS:
Biological: Tecemotide — Subjects who received tecemotide (L-BLP25) for the treatment of non-small cell lung cancer (NSCLC) or multiple myeloma in a feeder trial will continue to be treated with tecemotide (L-BLP25) and have safety assessments performed until the discontinuation criteria in the respective feeder trial protocol are met.
  Other Names: L-BLP25
  Arms: Tecemotide (L-BLP25)
Other: No intervention — Subjects who had not received tecemotide in the feeder study, or who had discontinued treatment with tecemotide (L-BLP25), will only be observed for progressive disease (PD) (if applicable) and survival in 6-month intervals and will not be provided treatment with tecemotide (L-BLP25).
  Arms: Observational

SUMMARY:
This is an open-label, common follow-up trial. Subjects who were enrolled in a Merck KGaA, EMD Serono or Merck Serono Japan sponsored trial with tecemotide (L-BLP25) were enrolled in this follow-up trial to continue their maintenance treatment with tecemotide (L-BLP25). Subjects were transferred once the feeder trial (EMR 63325-005 [NCT00157209], EMR 63325-006 [NCT00157196] and EMR 63325-008 [NCT01094548]) objectives were met. Subjects who received tecemotide (L-BLP25) in a feeder trial continued tecemotide (L-BLP25) treatment in this follow-up trial and have safety assessments performed as well as were observed for progressive disease (PD) and survival in 6- month intervals. Subjects who had not received tecemotide (L-BLP25) in feeder trials, or discontinued treatment were only observed for PD and survival in 6-month intervals and were not provided treatment with tecemotide (L-BLP25).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Registration and treatment in a clinical trial with tecemotide (L-BLP25) under sponsorship of Merck KGaA/EMD Serono/Merck Serono Japan (feeder trial). [Note, subjects who have been allocated to treatments not containing tecemotide (L BLP25) in the feeder trial are eligible for this trial and will be followed-up for progressive disease (PD) (if applicable) and survival.]
* End of Treatment procedures have been performed in the feeder trial.
* Other protocol defined inclusion criteria could apply

Exclusion Criteria

* Pregnancy and lactation period; women of childbearing potential, unless using effective contraception as determined by the Investigator. Subjects whom the Investigator considers may be at risk of pregnancy will have a pregnancy test performed per institutional standard
* Known hypersensitivity to any of the trial treatment ingredients (if applicable)
* Legal incapacity or limited legal capacity
* Any other reason that, in the opinion of the Investigator, precludes the subject from participating in the trial
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): January 2012/July 2012. Subjects randomized at 9 sites in Canada and Sweden.
Pre-assignment Details: Subjects who participated in the tecemotide (L-BLP25) clinical trials (EMR 63325-005, EMR 63325-006, and EMR 63325-008 served as feeder studies) were considered in this follow-up study after the protocol specific inclusion and exclusion criteria to continue their maintenance treatment. A total of 27 subjects were enrolled in this follow-up study.
Groups:
- Non-small Cell Lung Cancer (NSCLC); Multiple Myeloma: Subjects who received tecemotide in a feeder study continued treatment with tecemotide and had safety assessments performed until the discontinuation criteria described in the respective feeder study protocol were met. Once the subject discontinued maintenance treatment, an End of Treatment visit was performed. Thereafter, the subjects were observed for progression of disease (PD) (if applicable according to the respective feeder study protocol) and survival in 6-month intervals. Subjects who had not received tecemotide in the feeder study, or who had discontinued treatment with tecemotide, were only observed for PD (if applicable) and survival in 6-month intervals and were not provided treatment with tecemotide.
Period: Overall Study
Arm/Group | Non-small Cell Lung Cancer (NSCLC) | Multiple Myeloma
Started | 14 | 13
Number of Tecemotide Subjects | 12 | 8
Number of Non-treatment Subjects | 2 | 5
Safety Analysis Set | 12 | 8
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Screening analysis set included all the subjects included in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-small Cell Lung Cancer (NSCLC) | Multiple Myeloma | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (8.98) | 65.2 (9.81) | 66.5 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs), Serious AEs, AEs Leading to Discontinuation and AEs Leading to Death
Description: An Adverse Event (AE) is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A Serious AE is an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect, AEs leading to discontinuation and AEs leading to death.
Time Frame: Screening up to 42 days after last dose of study treatment with tecemotide (L-BLP25), assessed up to 3.6 years
Population: Only subjects treated with tecemotide were included in the safety analysis set.
Measure: Number; unit: Subjects
Groups:
- Non-small Cell Lung Cancer (NSCLC); Multiple Myeloma: Subjects who received tecemotide in a feeder study continued treatment with tecemotide and had safety assessments performed until the discontinuation criteria described in the respective feeder study protocol were met. Once the subject discontinued maintenance treatment, an End of Treatment visit was performed. Thereafter, the subjects were observed for progression of disease (PD) (if applicable according to the respective feeder study protocol) and survival in 6-month intervals.
Arm/Group | Non-small Cell Lung Cancer (NSCLC) | Multiple Myeloma
Number analyzed (Participants) | 12 | 8
Subjects
  AEs | 12 | 7
  Serious AE | 8 | 0
  AE leading to discontinuation | 2 | 0
  AE leading to death | 3 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival time was defined as the time from randomization to death. Subjects without events were censored at the last date they were known to be alive.
Time Frame: From randomization to death, assessed up to 3.6 years
Population: Efficacy analysis was not performed due to the premature termination of this safety follow-up study and the tecemotide program based on negative results in EMR 63325-009 (NCT00960115)
Arm/Group | Non-small Cell Lung Cancer (NSCLC) | Multiple Myeloma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening up to 42 days after last dose of study treatment with tecemotide (L-BLP25), assessed up to 3.6 years. AEs were reported only for Subjects who received tecemotide (L-BLP25) in feeder trial. No AEs were collected and reported for subjects who had not received tecemotide in the feeder study, or who had discontinued treatment with tecemotide (L-BLP25)
Groups:
- NSCLC; Multiple Myeloma: Subjects who received tecemotide in a feeder study continued treatment with tecemotide and had safety assessments performed until the discontinuation criteria described in the respective feeder study protocol were met. Once the subject discontinued maintenance treatment, an End of Treatment visit was performed. Thereafter, the subjects were observed for progression of disease (PD) (if applicable according to the respective feeder study protocol) and survival in 6-month intervals.
Arm/Group | NSCLC | Multiple Myeloma
Serious Adverse Events (participants affected / at risk) | 8/12 | 0/8
Other Adverse Events (participants affected / at risk) | 12/12 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC (N=12) | Multiple Myeloma (N=8)
Pneumonia (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC (N=12) | Multiple Myeloma (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0
Cataract (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 8 | 0
Influenza like illness (General disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 0
Injection site hypersensitivity (General disorders) | 1 | 0
Injection site induration (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 1
Oral allergy syndrome (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Infection parasitic (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 1
Lip infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Mycobacterial infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Onychomycosis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 5
Urinary tract infection (Infections and infestations) | 2 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 | 0
Radiation fibrosis (Injury, poisoning and procedural complications) | 1 | 0
Radiation fibrosis - lung (Injury, poisoning and procedural complications) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 1 | 0
Weight increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 5 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 2
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely as the sponsor decided to discontinue program with Tecemotide in non-small cell lung cancer (NSCLC).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator will inform the Sponsor in advance about any plans to publish or present data from the trial. Any publications and presentations of the results (abstracts in journals or newspapers, oral presentations, etc.), either in whole or in part, by Investigators or their representatives will require pre-submission review by the Sponsor.The Sponsor will not suppress or veto publications, but maintains the right to delay publication in order to protect intellectual property rights.